CLINICAL TRIAL: NCT01393431
Title: Exhaled Breath Condensate pH in Mechanically Ventilated Patients
Brief Title: Futility of Exhaled Breath Condensate pH Measurements in Ventilated Patients in Intensive Care Unit (ICU)
Status: Terminated | Type: Observational
Why Stopped: IRB recommended to stop the trial becasue none of the 4 procedures showed a predictive value for VAP, duration of MV or mortality.
Sponsor: Universidad Nacional de Rosario (Other)
Responsible Party: Luis J Nannini= Principal Investigator, Hospital Escuela E Perón & UNR
Other Study IDs: EBC pH in ICU
Record Dates: First submitted 2011-07-01; First posted 2011-07-13 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2008-05

CONDITIONS: Ventilator Associated Pneumonia; Death
Keywords: Exhaled breath condensate pH; Predictive value of pH
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EBC pH: Observational study

SUMMARY:
Measurement of pH in Exhaled breath condensate has been mentioned as a robust variable from lung inflammation. It is non-invasive and reproducible. The investigators measured pH in the water condensed in the trap of expiratory arm of ventilator.In ICU the investigators measured pH in condensed water without interfering with patients treatment. A group of critically ill patients mechanically ventilated due to non pulmonary cause were followed until successful weaning, death or pneumonia. The investigators found that pH did not change along the study and it did not predict worsening condition.

DETAILED DESCRIPTION:
Collection of exhaled breath condensate (EBC) became a promising method for obtaining samples from the lungs. In this prospective clinical trial we aimed to answer if spontaneous EBC in the trap of the expiratory arm of the ventilator could replace EBC collected by coolant chamber with gas standardization with Argon as an inert gas. Second, if EBC pH could predict ventilator associated pneumonia (VAP) and mortality. We included a group of critically ill patients, that required mechanical ventilation due to non-pulmonary cause. The patients were followed up until development of VAP, successful weaning or death.EBC pH spontaneously collected in the trap of expiratory arm of the ventilator. We measured pH with a blood gas analyzer, named Radiometer ABL5 Copenhagen. For the coolant chamber EBC pH measurement, the expiratory arm was passed through the chamber at -3ºC and in 10 min at least 2 ml was collected. The rest of the EBC was collected in Ependorff tube and pH was measured after de-aeration of the condensate with argon (350 ml/min) for 10 min as a gas standardization procedure as previously described by Hunt and colleagues. [Hunt JF, Fang K, Malik R, Snyder A, Malhotra N, Platts-Mills TAE, Gaston B. Endogenous airway acidification: implications for asthma pathophysiology. Am J Resp Crit Care Med 2000; 161: 694-699. ]

ELIGIBILITY:
Inclusion Criteria:

* Endotracheal intubation and mechanical ventilation for at least 48 hours due to non-pulmonary cause
* For whom their close acquaintances gave the informed consent

Exclusion Criteria:

* Pregnancy, denied surrogate decision-makers to give informed consent.
* Patients that required mechanical ventilation due to: pneumonia, severe respiratory infection, massive haemoptysis, acute severe asthma, bronchiectasis, COPD exacerbation, or acute lung injury. Finally, patients that expected to be ventilated less than 2 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (age >18) Acute critically ill patients that required endotracheal intubation and mechanical ventilation for at least 48 hours due to a non-pulmonary cause.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Exhaled Breath Condensate (EBC)pH of expiratory trap and Exhaled breath condensate pH obtained with coolant chamber and deaerated with Argon | follow up during mechanical ventilation, averaged less than 4 weeks
  It was an observational study that showed no changes in EBC pH despite different patient´s outcome. We, as investigators, did not make any intervention.

SECONDARY OUTCOMES:
Exhaled breath condensate pH could predict ventilator associated pneumonia or death | Follow up during mechanical ventilation (averaged less than 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Luis J Nannini, MD, Principal Investigator — hospital E Perón. UNR. ARGENTINA
Locations (1):
- Unidad de Terapia Intensiva. II Cátedra de Clínica Médica y Terapéutica. Universidad Nacional de Rosario. Hospital Escuela "Eva Perón". San Martín 1645., Granadero Baigorria, Santa Fe Province, Argentina